CLINICAL TRIAL: NCT06585020
Title: Amikacin Liposome Inhalation Suspension for Treatment of Mycobacterium Xenopi Pulmonary Infection
Acronym: AKAPI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Angers (Other Government); Hospital Avicenne (Other); University Hospital, Bordeaux (Other); University Hospital, Brest (Other); CH Compiègne (Unknown); Créteil Hospital (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Grenoble (Other); Centre Hospitalier le Mans (Other); Hôpital de la Croix-Rousse (Other); APHM - Nord (Unknown); Hôpital Saint Joseph (Unknown); CH Mulhouse (Unknown); CH Orléans (Unknown); Tenon Hospital, Paris (Other); Hôpital Necker-Enfants Malades (Other); Centre hospitalier de Perpignan (Other); Poitiers University Hospital (Other); CH Pontoise (Unknown); CHU de Reims (Other); Rennes University Hospital (Other); CHU de Rouen - Accueil (Other); Central Hospital Saint Quentin (Other Government); IHU Strasbourg (Other); University Hospital, Tours (Other); CH Abbeville (Unknown); CH Cannes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI2021_843_0148
Record Dates: First submitted 2024-08-13; First posted 2024-09-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Mycobacterium; Xenopi; Lung Diseases
Keywords: Mycobacterium; Xenopi; Lung Diseases
MeSH Terms: conditions — Mycobacterium Infections; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARIKAYCE (Experimental): Experimental arm = ARIKAYCE® during 6 months in addition to standard treatment (duration determined with date of sputum conversion)
  Interventions: Drug: Arikayce
- Standard treatment (Active Comparator): Control arm = standard treatment Standard treatment = Rifampicin, ethambutol and clarithromycin
  Interventions: Drug: standard treatment

INTERVENTIONS:
Drug: Arikayce — Treatment regimens containing three molecules, rifampicin, ethambutol, and clarithromycin with ARIKAYCE® during the 6 first months of treatment. After having confirmed the presence of all inclusion criteria and the absence of all exclusion criteria, and after having obtained the patient's free and informed consent, the patient will be included and randomized to one of the treatment regimens.
  Arms: ARIKAYCE
Drug: standard treatment — treatment regimens containing three molecules, rifampicin, ethambutol, and clarithromycin during the 6 first months of treatment. After having confirmed the presence of all inclusion criteria and the absence of all exclusion criteria, and after having obtained the patient's free and informed consent, the patient will be included and randomized to one of the treatment regimens.
  Arms: Standard treatment

SUMMARY:
Treatment of Mycobacterium xenopi (MX) lung disease is not-well- tolerated and concerned a growing number of patients, especially with chronic pulmonary diseases or immunosuppression. The outcome of these patients is poor, and treatment is very long. Indeed, this duration is based on the date of sputum conversion. Treatment should be continued until 12 months after sputum conversion. In the vast majority patients have converted after 6 months of treatment, so a 18 months duration in total. Unfortunately, few data are available for MX, as it is rare in USA, but it is the second NTM isolated in France and concerns an increasing number of patients. As it is uncommon in USA, no clinical studies conducted by the pharmaceutical laboratory will be planned. In a murine model of MX infection, the only drug which decreased the number colony formant units in mice lungs, was amikacin. Until now, amikacin was only available intravenously and used only for patients with very severe disease, because of renal and auditory toxicity. Amikacin liposome inhalation suspension (ARIKAYCE®) is amikacin sulfate encapsulated in liposomes for inhalational delivery. ARIKAYCE® increases amikacin uptake into alveolar macrophages, a refuge for NTM organisms; allows biofilm penetration; and limits systemic amikacin exposure ARIKAYCE® has already be tested in a randomized study on M. avium complex (MAC) refractory pulmonary infections. In this study, the culture conversion rate in the ARIKAYCE® group was higher than standard regimen group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* with an highly effective or acceptable contraception
* must present ATS/IDSA 2020 criteria for nontuberculous mycobacterial pulmonary infection
* the NTM should be M. xenopi

Exclusion Criteria:

* Patients presenting any of the following criteria cannot be included:
* Known hypersensitivity to one of the molecules of the study
* Relapse of MX lung infection
* Treatment with molecules able to interfere with cytochrome P450 that cannot be replaced by another therapeutic class
* HIV 1 and 2 human immunodeficiency virus infection
* Renal failure with creatinine clearance less than 30 mL/min
* Pregnancy and breastfeeding
* Cystic fibrosis
* Contraindications to one of the antibiotic :

Contraindication to the use of ARIKAYCE®:

* Hypersensitivity to the active substance, to aminoglycosides or to any of the excipients listed in section 6.1 of the CPR.
* Hypersensitivity to soy.
* Co-administration with any other aminoglycoside, regardless of the route of administration
* Severe Renal Failure

Contraindication to the use of Clarithromycine:

Allergy to macrolides or to any of the excipients listed in section 6.1;

* Association with :

  * colchicine,
  * ergot alkaloids, including for example dihydroergotamine, ergotamine, methylergometrine, methysergide: risk of ergotism,
  * pimozide, mizolastine: risk of QT interval prolongation and cardiac rhythm disorders, in particular ventricular tachycardia, ventricular fibrillation and torsades de pointes,
  * simvastatin, due to the increased risk of myopathy, including rhabdomyolysis.
  * lomitapide,
  * alfuzosin
  * dapoxetine
  * avanafil
  * ivabradine,
  * eplerenone,
  * dronedarone,
  * Quetiapine,
  * ticagrelor,
  * cisapride,
  * astemizole,
  * terfenadine,
  * ranolazine,
  * domperidone,
* Congenital or acquired prolongation of the QT interval (see sections 4.4 and 4.5 of the CPR)
* History of QT interval prolongation or ventricular rhythm disorders, in particular torsades de pointe (see sections 4.4 and 4.5 of the CPR);
* Electrolyte imbalances (hypokalaemia or hypomagnesaemia, due to the risk of QT interval prolongation) (see sections 4.4 and 4.5 of the CPR).Clarithromycin should not be used in patients with severe hepatic insufficiency in association with renal insufficiency.

Contraindication to the use of Rifampicine:

* Hypersensitivity to rifamycins or to any of the excipients listed in section 6.1 of the CPR.
* Porphyrias.
* Association with bictegravir, cobicistat, daclatasvir, dasabuvir, delamanid, grazoprevir/elbasvir, ritonavir-boosted protease inhibitors, isavuconazole, lédipasvir, lurasidone, midostaurine, ombitasvir/paritaprévir, praziquantel, rilpivirine, sofosbuvir, velpatasvir, voriconazole, voxilaprévir, (see section 4. 5 of the CPR). In children under 6 years of age, due to the risk of malaria

Contradiction the the use of Ethambutol:

* Known hypersensitivity to ethambutol
* Optic neuritis
* This medicine is contraindicated in patients with a wheat allergy (other than coeliac disease).
* Inability to comply with the requirements of the protocol, especially substance abuse, according to the investigator.
* Limited life expectancy (e.g 3 months)
* Patients with hematologic malignancies and allogeneic haematopoietic stem cells
* Women of childbearing age and not using an effective method of contraception (Pearl Index <1%)
* The patient is treated with molecules prolonging the QT interval that cannot be replaced by another therapeutic class.
* The patient presents a heart failure with left ventricular ejection fraction less than 30%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
variation of sputum conversion rate in ARIKAYCE® addition group compared to standard treatment | 3 months

SECONDARY OUTCOMES:
variation of time to culture conversion between both groups | at 3 month
variation of mortality between both groups | at 12 months
variation of mortality between both groups | at 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No